CLINICAL TRIAL: NCT00030043
Title: Penetrating Auditory Brainstem Implant for Neurofibromatosis 2
Brief Title: An Implant for Hearing Loss Due to Removal of Neurofibromatosis 2 Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: FD-R-001969-01
Record Dates: First submitted 2002-01-30; First posted 2002-01-31 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2002-01

CONDITIONS: Neurofibromatosis 2
Keywords: Electric Stimulation; Implants, Artificial; Brainstem; Electrodes; Speech Perception
MeSH Terms: conditions — Neurofibromatosis 2

INTERVENTIONS:
Device: Penetrating auditory brainstem implant

SUMMARY:
This is a study to gather some information on the safety and efficacy of the penetrating auditory brainstem implant (PABI) in patients with neurofibromatosis type 2.

DETAILED DESCRIPTION:
Neurofibromatosis Type 2 (NF2) is characterized by multiple tumors of the cranial and spinal nerves, and, in particular, by bilateral acoustic tumors. Surgical resection of these tumors generally results in the transection of the VIIIth nerve, destruction of the cochlea and auditory nerve, and total hearing loss. Due to the loss of the auditory nerve, these patients are not candidates for cochlear implantation. The Auditory Brainstem Implant (ABI) provides the only available intervention to restore some auditory sensation to these patients. An ABI is an implantable prosthesis that produces sound sensation by electrical stimulation of the ascending auditory pathway at the level of the cochlear nucleus.

The PABI may be placed surgically during tumor resection. Efficacy will be assessed using psychophysical and standard speech reception measures.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of neurofibromatosis type 2
* Speak English as a primary language

Exclusion criteria:

* Physical, psychological, or medical conditions that contraindicate the surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2001-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - House Ear Institute, Los Angeles, California
  - Huntington Medical Research Institutes, Pasadena, California
  - Cochlear Corporation, Englewood, Colorado